CLINICAL TRIAL: NCT03024632
Title: Trial of Labor After 3 or More Previous Cesarean Sections
Brief Title: Previous Cesarean Sections
Status: Withdrawn | Type: Observational
Why Stopped: Closed study. Study is retrospective in nature and never enrolled any subjects.
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Christopher Buchanan, MD, Principal Investigator, St. Louis University
Other Study IDs: 27685
Record Dates: First submitted 2017-01-13; First posted 2017-01-19 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Trial of Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- trial of labor: Pregnant women with a history of 3 or more cesarean sections who desired a trial of labor
  Interventions: Procedure: Trial of labor
- No trial of labor: Pregnant women with a history of 3 or more cesarean sections who desired a a repeat cesarean section

INTERVENTIONS:
Procedure: Trial of labor — trial of labor after 3 or more previous cesarean deliveries
  Groups: trial of labor

SUMMARY:
This is a retrospective chart review. The purpose is to look at the outcomes for women and newborns who decided to attempt a trial of labor after 3 or more previous cesarean sections.

DETAILED DESCRIPTION:
In 2006, the vaginal birth after cesarean (VBAC) rate was 8.5%, compared to a rate of 28.3% in 1996. This was also associated with a rise in the rate of cesarean section from approximately 20% to 31.1% over that same period of time. In that 10 year period, some hospitals stopped offering a trial of labor after cesarean (TOLAC) altogether.

Currently, the American College of Obstetricians and Gynecologists states in Practice Bulletin 115 (2010), Vaginal Birth After Previous Cesarean Delivery, "it is reasonable to consider women with 2 previous low transverse cesarean deliveries to be candidates for TOLAC…Data regarding the risk for women undergoing TOLAC with more than two previous cesarean deliveries is limited."

In 1994, a study reviewing10 years of data regarding trial of labor after cesarean. Of their population with 3 or more previous cesarean deliveries, 30% of patients underwent a trial of labor, with a 79% success rate. In this group, the uterine rupture rate was 1.2% with zero perinatal deaths related to rupture, which is compared to a rupture rate of 1.8% and 1 perinatal death in the group of 2 previous cesarean deliveries.

In 2002, another study described the outcomes of women who underwent a trial of labor after 2 or more previous cesarean deliveries at two large university hospitals in the Netherlands, but it included just 59 patients total and only 4 of these had 3 previous cesarean deliveries. No patients with more than 3 previous cesarean deliveries had a trial of labor.

A study in 2010, described a large cohort of women from the northeastern United States with 3 or more previous cesarean deliveries, including those attempting VBAC. This cohort included 89 women, of whom 79.8% had a successful VBAC. However, of the women who had a TOLAC, 40.4% delivered in a university hospital and only 18.0% in a hospital with an OB/GYN residency, compared to 56.9% and 25.4% of women who had an elective repeat cesarean section. In the group that had a TOLAC, there were no cases of uterine rupture.

There still remains a lack of data about the outcomes of the delivery of women who desire a trial of labor after 3 or more previous cesarean deliveries at a single institution.

The investigators will analyze and compare the management and outcomes of women and neonates for patients who attempted a trial of labor after 3 or more previous cesareans. We will also compare them to women and neonates of patients who underwent a repeat cesarean section without a trial of labor.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of 3 or more cesarean sections
* pregnant
* singleton

Exclusion Criteria:

* Less than 3 cesarean sections

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 14-55yrs of age Pregnant all ethnic backgrounds
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of Vaginal births | Labor through 6 weeks postpartum
  outcomes and safety of a trial of labor after 3 or more previous c-sections managed at a tertiary care facility

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Q Buchanan, MD, Study Director — St. Louis University

IPD SHARING:
Plan to Share IPD: No